CLINICAL TRIAL: NCT02399709
Title: Pilot Randomized Double Blind, Placebo Controlled Trial of the Efficacy of Simvastatin for Smoking Cessation
Brief Title: Trial to Evaluate the Efficacy of Simvastatin for Smoking Cessation
Acronym: ADDICSTATINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADDICSTATINE
Record Dates: First submitted 2015-03-20; First posted 2015-03-26 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- simvastatin (Experimental): oral administration, capsule of 20mg.
  Interventions: Drug: simvastatin
- microcrystalline cellulose (Placebo Comparator): oral administration, capsule of 20mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: simvastatin
  Arms: simvastatin
Drug: Placebo
  Arms: microcrystalline cellulose

SUMMARY:
Tobacco smoking is the number one preventable cause of disease worldwide. Unfortunately, there are few smoking cessation agents and their effectiveness has been shown to be relatively limited and is associated with potential unwanted effects. Therefore, the discovery of new medications that can facilitate abstinence and reduce relapse to cigarette use represents a pressing necessity. In the attempt to find molecules that could reduce drug-seeking behavior, we discovered that simvastatin reduces cocaine and nicotine, but not food, seeking behavior in rats. This discovery of a new therapeutic application for an already marketed class of compounds may greatly facilitate the translation from preclinical to clinical setting. In this project, we aim at investigating whether simvastatin is an effective smoking cessation agent in humans.

The study design is a multicenter, randomized, double blind 2 parallel groups, clinical trial with an intention-to-treat analysis. Smokers will randomly be assigned to receive simvastatin or placebo for 3 months. 200 smokers (100 receiving simvastatin and 100 receiving placebo) will be recruited through already established networks of general practitioners. The primary outcome of the efficacy of simvastatin will be the rate of smoking abstinence during the last month of the 3-month treatment period, defined as reported continuous abstinence from smoking and confirmed by expired air carbon monoxide and urinary cotinine concentration. The last assessment will be done 6 months after the predefined quit date.

The results of this proof-of-concept study may open new perspectives in the treatment of tobacco use and dependance.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 and <=70 years,
* Smoking more than 10 cigarettes per day for at least 1 year,
* Motivated to quit smoking,
* Without legal tutors or subordination,
* Affiliated to a health insurance system as required by the French law on biomedical research,
* Written informed consent for participation in the study.

Exclusion Criteria:

* Age < 18 or > 70 years,
* Presenting a contraindication to simvastatin use,
* With depression and/or psychosis and/or cognitive disorder and/or mental retardation or chronic use of medications for these disorders,
* Substance use disorder other than smoking,
* More than 3 months of abstinence from cigarette smoking in the previous year,
* Use of nicotine replacement therapy, bupropion, varenicline on last 3 months,
* Use of clonidine or nortriptyline on last 3 months,
* Undergoing on last 3 months' cognitive-behavioral therapy for smoking cessation,
* Premenopausal women without contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-10-08 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Self-reported number of cigarettes smoked | After 3 months of simvastatin treatment

SECONDARY OUTCOMES:
Self-reported continuous abstinence during the last 4 weeks of the 3 months of treatment with simvastatin versus placebo | After 3 months of simvastatin treatment
Expired air carbon monoxide ≤ 8 ppm | After 3 months of simvastatin treatment
Urinary cotinine concentration ≤ 10 ng/mL | After 3 months of simvastatin treatment
Nicotine craving assessed by the FTCQ-12 | After 3 months of simvastatin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine PERAULT-POCHAT, MD, PhD, Principal Investigator — Poitiers University Hospital
Locations (1):
- Poitiers University Hospital, Poitiers, France